CLINICAL TRIAL: NCT02509078
Title: Reevaluation Of Systemic Early Neuromuscular Blockade
Acronym: ROSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Boyd Taylor Thompson, Prinicipal Investigator PETAL CCC, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PETAL01ROSE; 1U01HL123009-01 (NIH)
Record Dates: First submitted 2015-07-24; First posted 2015-07-27 (Estimated); Results first posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-07

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ARDS; neuromuscular blocker; cisatracurium
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — cisatracurium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early Neuromuscular Blockade (NMB) (Active Comparator): Patients will receive cisatracurium besylate for the first 48 hours of the trial.
  Interventions: Drug: Cisatracurium Besylate
- Control: No Routine Early NMB (No Intervention): Use of non-study NMB will be discouraged.

INTERVENTIONS:
Drug: Cisatracurium Besylate — Patients randomized to the early neuromuscular blockade arm will receive a cisatracurium besylate bolus of 15 mg, followed by a continuous infusion of 37.5 mg/hour for 48 hours. Patients randomized to the control arm will receive no protocol specified neuromuscular blockade.
  Other Names: Nimbex
  Arms: Early Neuromuscular Blockade (NMB)

SUMMARY:
This study evaluates whether giving a neuromuscular blocker (skeletal muscle relaxant) to a patient with acute respiratory distress syndrome will improve survival. Half of the patients will receive a neuromuscular blocker for two days and in the other half the use of neuromuscular blockers will be discouraged.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

To assess the efficacy and safety of early neuromuscular blockade in reducing mortality and morbidity in patients with moderate-severe ARDS, in comparison to a control group with no routine early neuromuscular blockade (NMB).

PRIMARY HYPOTHESIS:

Early neuromuscular blockade will improve mortality prior to discharge home before day 90, in patients with moderate-severe ARDS.

The trial will accrue a maximum of 1408 patients. Patients will be recruited from the emergency departments, intensive care units and other acute care areas of the PETAL Network Clinical Centers and randomized to the active (NMB) or control. The overall strategy is to screen, consent, and enroll early, every newly intubated, acutely ill or post-operative, eligible patient at each site, using clinically obtained pulse oximetry and blood gases.

By preventing active expiration, and/or patient ventilator dyssynchrony, neuromuscular blockade may create a more homogenous distribution of airway pressures and tidal volumes, preventing barotrauma/volutrauma and "atelectrauma" resulting in less ventilator-induced lung injury.

ELIGIBILITY:
Inclusion Criteria

1. Age > 18 years
2. Presence of all of the following conditions for < 48 hours:

   i. PaO2/FiO2 < 150 with PEEP >/= 8 cm H2O OR, if ABG not available, SaO2/FiO2 ratio that is equivalent to a PaO2/FiO2 < 150 with PEEP >/= 8 cm H2O , and a confirmatory SaO2/FiO2 ratio that is again equivalent 1-6 hours later

ii. Bilateral opacities not fully explained by effusions, lobar/lung collapse, or nodules.

iii. Respiratory failure not fully explained by cardiac failure or fluid overload; need objective assessment (e.g., echocardiography) to exclude hydrostatic edema if no risk factor present.

Patients must be enrolled within 48 hours of meeting inclusion criteria.

Exclusion Criteria:

1. Lack of informed consent
2. Continuous neuromuscular blockade at enrollment
3. Known pregnancy
4. Currently receiving ECMO therapy
5. Chronic respiratory failure defined as PaCO2 > 60 mm Hg in the outpatient setting
6. Home mechanical ventilation (non-invasive ventilation or via tracheotomy) except for CPAP/BIPAP used solely for sleep-disordered breathing
7. Actual body weight exceeding 1 kg per centimeter of height
8. Severe chronic liver disease defined as a Child-Pugh score of 12-15 (Appendix A2)
9. Bone marrow transplantation within the last 1 year
10. Expected duration of mechanical ventilation of < 48 hours
11. Decision to withhold life-sustaining treatment; except in those patients committed to full support except cardiopulmonary resuscitation if an actual cardiac arrest occurs
12. Moribund patient not expected to survive 24 hours; if CPR provided, assess for moribund status greater than 6 from CPR conclusion
13. Diffuse alveolar hemorrhage from vasculitis
14. Burns > 70% total body surface
15. Unwillingness to utilize the ARDS Network 6 ml/kg IBW ventilation protocol
16. Previous hypersensitivity or anaphylactic reaction to cisatracurium
17. Neuromuscular conditions that may potentiate neuromuscular blockade and/or impair spontaneous ventilation (Appendix A2)
18. Neurologic conditions undergoing treatment for intracranial hypertension
19. Enrollment in an interventional ARDS trial with direct impact on neuromuscular blockade and PEEP
20. >120 hours of mechanical ventilation
21. P/F < 200 mmHg at the time of randomization (if available)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1008 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2018-07-03 (Actual); Study Completion 2019-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A. Schoenfeld, PhD, Principal Investigator — Massachusetts General Hospital
Locations (44):
- United States (44):
  - UCSF Fresno, Fresno, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - UCSF Medical Center, San Francisco, California
  - Stanford University Hospital, Stanford, California
  - Medical Center of Aurora, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Indiana University Methodist Hospital, Indianapolis, Indiana
  - University Medical Center, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - St. Vincent's Hospital, Worcester, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Henry Ford Medical Center, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Mt. Sinai Hospital, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Wesley Long Hospital, Greensboro, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Summa Akron City Hospital, Akron, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - UPMC Presbyterian/Mercy/Shadyside, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - University Hospital, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - University or Virginia Health System, Charlottesville, Virginia
  - VCU Medical Center, Richmond, Virginia
  - Harborview Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Swedish Hospital Cherry Hill, Seattle, Washington
  - Swedish Hospital First Hill, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Data will be collected electronically and stored at the Clinical Coordinating Center at MGH. A de-identified database of all data will be available for use 3 years after the primary publication. Data can be accessed at that point via the NHLBI BioLINCC data repository.

REFERENCES:
- [Derived] National Heart, Lung, and Blood Institute PETAL Clinical Trials Network; Moss M, Huang DT, Brower RG, Ferguson ND, Ginde AA, Gong MN, Grissom CK, Gundel S, Hayden D, Hite RD, Hou PC, Hough CL, Iwashyna TJ, Khan A, Liu KD, Talmor D, Thompson BT, Ulysse CA, Yealy DM, Angus DC. Early Neuromuscular Blockade in the Acute Respiratory Distress Syndrome. N Engl J Med. 2019 May 23;380(21):1997-2008. doi: 10.1056/NEJMoa1901686. Epub 2019 May 19. PMID 31112383
- [Derived] Sjoding MW, Schoenfeld DA, Brown SM, Hough CL, Yealy DM, Moss M, Angus DC, Iwashyna TJ; NHLBI Prevention and Early Treatment of Acute Lung Injury (PETAL) Network. Power Calculations to Select Instruments for Clinical Trial Secondary Endpoints. A Case Study of Instrument Selection for Post-Traumatic Stress Symptoms in Subjects with Acute Respiratory Distress Syndrome. Ann Am Thorac Soc. 2017 Jan;14(1):110-117. doi: 10.1513/AnnalsATS.201608-585OC. PMID 27788018
- [Derived] Huang DT, Angus DC, Moss M, Thompson BT, Ferguson ND, Ginde A, Gong MN, Gundel S, Hayden DL, Hite RD, Hou PC, Hough CL, Iwashyna TJ, Liu KD, Talmor DS, Yealy DM; Reevaluation of Systemic Early Neuromuscular Blockade Protocol Committee and the National Institutes of Health National Heart, Lung, and Blood Institute Prevention and Early Treatment of Acute Lung Injury Network Investigators. Design and Rationale of the Reevaluation of Systemic Early Neuromuscular Blockade Trial for Acute Respiratory Distress Syndrome. Ann Am Thorac Soc. 2017 Jan;14(1):124-133. doi: 10.1513/AnnalsATS.201608-629OT. PMID 27779896
- See also: Website for the PETAL Network — http://petalnet.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: No Routine Early NMB: Use of non-study NMB will be discouraged. Patients randomized to the control arm will receive no protocol specified neuromuscular blockade.
Period: Overall Study
Arm/Group | Early Neuromuscular Blockade (NMB) | Control: No Routine Early NMB
Started | 502 | 506
Completed | 501 | 505
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Neuromuscular Blockade (NMB) | Control: No Routine Early NMB | Total
Number analyzed (Participants) | 501 | 505 | 1006
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 348 | 358 | 706
  >=65 years | 153 | 147 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (14.7) | 55.1 (15.9) | 55.8 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 210 | 236 | 446
  Male | 291 | 269 | 560
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 64 | 54 | 118
  Not Hispanic or Latino | 410 | 421 | 831
  Unknown or Not Reported | 27 | 30 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 3 | 8
  Asian | 10 | 10 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 61 | 79 | 140
  White | 360 | 343 | 703
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 63 | 69 | 132
Region of Enrollment [Number; unit: participants]
  United States | 501 | 505 | 1006

OUTCOME MEASURES:

1. Primary Outcome: Hospital Mortality to Day 90
Description: The percentage of subjects alive at study day 90. Those subjects discharged home prior to day 90 were counted as alive at day 90.
Time Frame: 90 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Early Neuromuscular Blockade (NMB) | Control: No Routine Early NMB
Number analyzed (Participants) | 501 | 505
Participants
  Alive at Day 90 | 288 | 289
  Dead Prior to Day 90 | 213 | 216
Statistical Analysis 1: Comparison: Early Neuromuscular Blockade (NMB) vs Control: No Routine Early NMB; Test type: Superiority; p = 0.93, Wald test for the difference of two prop; Risk Difference (RD) = -0.3, 95% CI 2-sided [-6.4 to 5.9] — Estimated value is a percentage

2. Secondary Outcome: Mean Ventilator Free Days to Day 28
Description: Ventilator-free days is defined to be 28 days minus the duration of mechanical ventilation through day 28. Participants who do not survive to day 28 are assigned zero ventilator-free days.
Time Frame: 28 days after randomization
Population: The overall number of participants analyzed reflects the number of patients that had sufficient data to allow for calculation of the outcome measure.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Early Neuromuscular Blockade (NMB) | Control: No Routine Early NMB
Number analyzed (Participants) | 500 | 505
days | 9.6 (10.4) | 9.9 (10.9)

3. Secondary Outcome: Mean Organ Failure Free Days to Day 28
Description: SOFA (Sepsis-related Organ Failure Assessment) was used to determine criteria for an organ failure free day. Scores were based on four of the six SOFA organ categories: Coagulation, Liver, Cardiovascular, and Renal. Each category was scored 0-4; 0 being normal functioning and 4 being the most abnormal. A patient was considered failure free on each day alive with SOFA scores below 2 for all four organ systems.
  Ref: Vincent, J.L., et al., The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med, 1996. 22(7): p. 707-10.
Time Frame: 28 days after randomization
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Early Neuromuscular Blockade (NMB) | Control: No Routine Early NMB
Number analyzed (Participants) | 480 | 479
days | 12.4 (11.3) | 12.5 (11.5)

4. Secondary Outcome: ICU Free Days to Day 28
Description: ICU free days is defined as the number of days between randomization and day 28 in which the patient is in the ICU (for any part of a day).
Time Frame: 28 days after randomization
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Early Neuromuscular Blockade (NMB) | Control: No Routine Early NMB
Number analyzed (Participants) | 500 | 505
days | 9.0 (9.4) | 9.4 (9.8)

5. Secondary Outcome: Mean Hospital Free Days to Days 28
Description: Hospital free days are days alive post hospital discharge through day 28. Patients who die on or prior to day 28 are assigned zero hospital free days.
Time Frame: 28 days after randomization
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Early Neuromuscular Blockade (NMB) | Control: No Routine Early NMB
Number analyzed (Participants) | 501 | 505
days | 5.7 (7.8) | 5.9 (8.1)

6. Secondary Outcome: Katz Activities of Daily Living (ADL)/Lawton Instrumental Activities Of Daily Living Scale (IADL)
Description: Assesses whether individual can living independently and assess a range of common functional activities, from walking and toileting to managing money and cooking meals. Data is a pooled estimates from patient survey and proxy survey. The total score is rated from 0 to 10 (MCID=1; 1 point=1 ADL); a higher score indicates having more difficulties in daily activities.
Time Frame: 3 months after randomization
Population: The overall number of participants analyzed reflects the number of patients that were alive, able to be contacted, and had sufficient data to allow for calculation of the outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Early Neuromuscular Blockade (NMB) | Control: No Routine Early NMB
Number analyzed (Participants) | 212 | 196
score on a scale | 3.3 (2.7) | 3.0 (2.7)

7. Secondary Outcome: EuroQol (EQ-5D-5L): Health Related Quality of Life
Description: Using a standardized scale, do health reasons limit the person's ability to enjoy their life? Pooled estimates from patient survey and proxy survey were used. Utility index was computed from a lookup table according to EQ-5D-5L response profiles; utility index ranges from -0.11 to 1.00 (higher scores are better; 1.00 is perfect health), minimal clinically important difference (MCID) is 0.07
Time Frame: 3 months after randomization
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Early Neuromuscular Blockade (NMB) | Control: No Routine Early NMB
Number analyzed (Participants) | 207 | 194
score on a scale | 0.66 [0.41 to 0.82] | 0.73 [0.44 to 0.83]

8. Secondary Outcome: PTSS-14: Post-traumatic Stress-like Symptoms Scores >/= 45
Description: Does the patient have symptoms of anxiety and stress from their ICU stay? PTSS-14 is only asked at month 6 and month 12 in patient survey; total score is rated from 14 to 98 and a higher score indicates having more post-traumatic stress syndrome related symptoms. Participants with scores greater than or equal to 45 were reported.
Time Frame: 6 months after randomization
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Early Neuromuscular Blockade (NMB) | Control: No Routine Early NMB
Number analyzed (Participants) | 145 | 122
participants | 38 | 31

9. Secondary Outcome: MoCA-Blind: Montreal Cognitive Assessment
Description: How clearly can patient think and recall things? MoCA-Blind is only asked in patient survey; total score is rated from 0 to 30 and a higher score indicates better cognitive performance. Normal range: 26 or greater.
Time Frame: 3 months after randomization
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Early Neuromuscular Blockade (NMB) | Control: No Routine Early NMB
Number analyzed (Participants) | 154 | 133
score on a scale | 22.2 (5.2) | 22.8 (4.8)

10. Secondary Outcome: Katz Activities of Daily Living (ADL)/Lawton Instrumental Activities Of Daily Living Scale (IADL)
Description: as for outcome 6
Time Frame: 6 months after randomization
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Early Neuromuscular Blockade (NMB) | Control: No Routine Early NMB
Number analyzed (Participants) | 180 | 156
score on a scale | 2.7 (2.4) | 2.7 (2.4)

11. Secondary Outcome: Katz Activities of Daily Living (ADL)/Lawton Instrumental Activities Of Daily Living Scale (IADL)
Description: as for outcome 6
Time Frame: 12 months after randomization
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Early Neuromuscular Blockade (NMB): Patients will receive cisastracurium besylate for the first 48 hours of the trial.
  cisastracurium besylate: Patients randomized to the early neuromuscular blockade arm will receive a cisastracurium besylate bolus of 15 mg, followed by a continuous infusion of 37.5 mg/hour for 48 hours. Patients randomized to the control arm will receive no protocol specified neuromuscular blockade.
Arm/Group | Early Neuromuscular Blockade (NMB) | Control: No Routine Early NMB
Number analyzed (Participants) | 128 | 119
score on a scale | 2.9 (2.6) | 2.4 (2.3)

12. Secondary Outcome: EuroQol (EQ-5D-5L): Health Related Quality of Life
Description: as for outcome 7
Time Frame: 6 months after randomization
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Early Neuromuscular Blockade (NMB) | Control: No Routine Early NMB
Number analyzed (Participants) | 176 | 155
score on a scale | 0.74 [0.57 to 0.83] | 0.79 [0.55 to 0.83]

13. Secondary Outcome: EuroQol (EQ-5D-5L): Health Related Quality of Life
Description: as for outcome 7
Time Frame: 12 months after randomization
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Early Neuromuscular Blockade (NMB) | Control: No Routine Early NMB
Number analyzed (Participants) | 127 | 119
score on a scale | 0.75 [0.57 to 0.83] | 0.77 [0.57 to 0.86]

14. Secondary Outcome: MoCA-Blind: Montreal Cognitive Assessment
Description: as for outcome 9
Time Frame: 6 months after randomization
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Early Neuromuscular Blockade (NMB) | Control: No Routine Early NMB
Number analyzed (Participants) | 138 | 114
score on a scale | 22.8 (4.8) | 23.2 (5.1)

15. Secondary Outcome: MoCA-Blind: Montreal Cognitive Assessment
Description: as for outcome 9
Time Frame: 12 months after randomization
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Early Neuromuscular Blockade (NMB) | Control: No Routine Early NMB
Number analyzed (Participants) | 99 | 88
score on a scale | 23.3 (4.9) | 24.0 (4.4)

16. Secondary Outcome: PTSS-14: Post-traumatic Stress-like Symptoms Scores >/= 45
Description: as for outcome 8
Time Frame: 12 months after randomization
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Early Neuromuscular Blockade (NMB) | Control: No Routine Early NMB
Number analyzed (Participants) | 103 | 94
participants | 21 | 38

ADVERSE EVENTS:
Time Frame: Subjects were assessed for occurrence of adverse events from time of randomization through study day 7 (five days after infusion of study drug) or ICU discharge, whichever occurred first.
Arm/Group | Early Neuromuscular Blockade (NMB) | Control: No Routine Early NMB
All-Cause Mortality (participants affected / at risk) | 213/501 | 216/505
Serious Adverse Events (participants affected / at risk) | 28/501 | 21/505
Other Adverse Events (participants affected / at risk) | 19/501 | 15/505
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Early Neuromuscular Blockade (NMB) (N=501) | Control: No Routine Early NMB (N=505)
Methemoglobinemia (Blood and lymphatic system disorders) | 1 | 0
AV Block complete (Cardiac disorders) | 1 | 0
Atrial Fibrillation with RVR (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 6 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0
Tachycardia Supraventricular (Cardiac disorders) | 1 | 0
Torsades De Pointe (Cardiac disorders) | 1 | 0
Ventricular Tachycardia (Cardiac disorders) | 2 | 0
Death (General disorders) | 1 | 0
Necrosis of left foot (General disorders) | 1 | 0
Reaction Febrile (General disorders) | 1 | 0
Cerebral Infartion (Nervous system disorders) | 1 | 0
CVA (Nervous system disorders) | 1 | 0
Hemmorage Brain (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Stroke (Nervous system disorders) | 3 | 0
Subdural Effusion (Nervous system disorders) | 1 | 0
Airway Obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Embolus Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laceration Diaphragm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hypotension (Vascular disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 2
Heart Block Av 3rd Degree (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Bleeding Intracranial (Nervous system disorders) | 0 | 1
Cerebral Infarction (Nervous system disorders) | 0 | 1
Hemorrhage Brain (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 1
Stroke (Nervous system disorders) | 0 | 1
Subarachnoid Hemorrhage (Nervous system disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Hematoma (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Early Neuromuscular Blockade (NMB) (N=501) | Control: No Routine Early NMB (N=505)
Atrial Fibrillation Paroxysmal (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac Arrhythmia (Nos) (Cardiac disorders) | 1 | 0
Severe Prolonged Bradycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Paralysis Awareness (Injury, poisoning and procedural complications) | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Subcutaneous Emphysema And Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 6 | 0
Superficial Venous Thrombus (Vascular disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 2
Vasovagal Reaction (Cardiac disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Stoma Leak (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hemorrhage Retroperitoneal (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In addition to the restriction on the PI for sponsor to review results prior to public release within 60 days, there is a network provision: The Publications Committee of the PETAL Network must review and approve all pre-submission PETAL Network studies before publication or presentation. Manuscripts comparing outcomes of PETAL study endpoints from one center to the reminder of the group are not permitted.

DOCUMENTS (2):
  • Study Protocol (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/78/NCT02509078/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/78/NCT02509078/SAP_001.pdf